CLINICAL TRIAL: NCT04345367
Title: A PHASE 3B RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY, ACTIVE CONTROLLED MULTI-CENTER STUDY ASSESSING THE EFFICACY AND SAFETY OF ABROCITINIB COMPARED WITH DUPILUMAB IN ADULT PARTICIPANTS ON BACKGROUND TOPICAL THERAPY WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study of Abrocitinib Compared With Dupilumab in Adults With Moderate to Severe Atopic Dermatitis on Background Topical Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451050; 2019-004013-13 (EudraCT Number)
Record Dates: First submitted 2020-03-27; First posted 2020-04-14 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib; dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Abrocitinib 200 mg plus placebo injection (Experimental): Abrocitinib 200 mg daily through Week 26, plus placebo injections every other week through Week 24
  Interventions: Drug: Abrocitinib 200 mg
- Dupilumab 300 mg plus placebo tablets (Active Comparator): Dupilumab 300 mg every other week (2 injections on Day 1) through Week 24, plus placebo tablets daily through Week 26
  Interventions: Combination Product: Dupilumab 300 mg

INTERVENTIONS:
Drug: Abrocitinib 200 mg — Abrocitinib 200 mg administered as two 100 mg tablets to be taken orally once daily for 26 weeks. Placebo injections will be administered every other week for 24 weeks.
  Arms: Abrocitinib 200 mg plus placebo injection
Combination Product: Dupilumab 300 mg — Dupilumab 300 mg administered as a single subcutaneous injection every other week for 24 weeks (2 injections on day 1). Placebo tablets will be administered daily.
  Arms: Dupilumab 300 mg plus placebo tablets

SUMMARY:
This is a randomized, double-blind, double-dummy, active-controlled, multi-center study to assess the efficacy and safety of abrocitinib 200 mg (2 x 100 mg tablets) administered orally QD compared with dupilumab 300 mg administered by subcutaneous injection every other week (as per label guidelines) in adult participants on background topical therapy, with moderate to severe AD. The treatment duration is 26 weeks. A total of approximately 600 participants will be enrolled from approximately 220 sites globally. Approximately 600 participants will be randomly assigned to study intervention. There are primary efficacy assessments at Week 2 and Week 4, and a key secondary efficacy assessment at Week 16. Efficacy and safety endpoints will be assessed throughout the entire study. Exploratory endpoints related to hand eczema efficacy will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of chronic atopic dermatitis (AD) for at least 6 months
* Moderate to severe AD (BSA at least 10%, IGA at least 3, EASI at least 16, and PP-NRS severity score at least 4)
* Recent history of inadequate response to treatment with medicated topical therapy for AD, or who have required systemic therapies for control of their disease

Exclusion Criteria:

* Acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation
* Have increased risk of developing venous thromboembolism
* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Prior treatment with systemic JAK inhibitors or IL-4 or IL-13 antagonists including dupilumab, lebrikizumab or tralokinumab
* Other active non-AD inflammatory skin diseases or conditions affecting skin
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, malignancies, current or history of certain infections, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (151):
- United States (49):
  - Total Skin & Beauty Dermatology Center, PC, Birmingham, Alabama
  - Clinical Research Center Of Alabama, Birmingham, Alabama
  - Alliance Dermatology & MOHS Center, PC, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Ark Clinical Research, Long Beach, California
  - Beach Allergy and Asthma Specialty Group, A Medical Corporation, Long Beach, California
  - Wallace Medical Group, Inc, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - MedDerm Associates, San Diego, California
  - University of California San Diego Dermatology, San Diego, California
  - University Clinical Trials Inc., San Diego, California
  - Synergy Dermatology, San Francisco, California
  - Wolverine Clinical Trials, Llc, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Skin Care Research, LLC, Boca Raton, Florida
  - Olympian Clinical Research, Largo, Florida
  - Miami Dermatology & Laser Research, LLC, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Accel Research Sites - Pure Skin Dermatology & Aesthetics, Orlando, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Integrated Clinical Research, West Palm Beach, Florida
  - One Health Research Clinic, Norcross, Georgia
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Avant Research Associates, LLC, Crowley, Louisiana
  - MetroBoston Clinical Partners, LLC, Brighton, Massachusetts
  - Onyx Clinical Research, Flint, Michigan
  - Linden Road Imaging Center, Flint, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Regional Medical Imaging, P.C. ( Local X-Ray), Royal Oak, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Skin Specialists, PC, Omaha, Nebraska
  - Vivida Dermatology, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Boice-Willis Clinic, PA, Rocky Mount, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Acclaim Dermatology, PLLC, Sugar Land, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah
- Australia (8):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Melbourne Health Radiology, Pakrville, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (5):
  - MHAT Dobrich AD, Dobrich
  - MC Asklepii OOD, Dupnitsa
  - DCC Alexandrovska EOOD, Sofia
  - DCC Fokus-5 - Medical Establishment for Outpatient Care EOOD, Sofia
  - Military Medical Academy MHAT Sofia, Sofia
- Canada (21):
  - Dermatology Research Institute, Calgary, Alberta
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - CARE Clinic Ltd, Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Karma Clinical Trials, Inc., St. John's, Newfoundland and Labrador
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Intermed groupe santé, Chicoutimi, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Chile (8):
  - Medicien, Las Condes, Santiago, Santiago Metropolitan
  - MIRES (M Y F Estudios Clinicos Limitada), Nunoa, Santiago, Santiago Metropolitan
  - Vida lntegra, Nunoa, Santiago, Santiago Metropolitan
  - Centro Radiologico Plaza Baquedano, Santiago, Santiago Metropolitan
  - Centro Medico SkinMed Limitada, Santiago, Santiago Metropolitan
  - Clínica Dermacross S.A., Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
- Finland (3):
  - Terveystalo Tampere, Tampere
  - Mehiläinen Neo, Turku
  - Turun yliopistollinen keskussairaala, Turku
- Germany (10):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Klinikum Bielefeld Rosenhöhe, Bielefeld
  - Klinische Forschung Dresden GmbH, Dresden
  - IKF Pneumologie GmbH & Co KG, Frankfurt am Main
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Studienzentrum Dr. med. Beate Schwarz, Langenau
  - SIBAmed GmbH, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - University of Muenster, Münster
- Hungary (4):
  - Clinexpert Kft., Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Trial Pharma Kft., Kaposvár
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Fondazione Policlinico Universitario A. Gemelli IRCCS Universita Cattolica del Sacro Cuore, Roma, Italy
- Latvia (3):
  - Health Centre 4 Ltd. Diagnostics Centre, Riga
  - LLC J.Kisis, Riga
  - Outpatient Clinic of Ventspils, Ventspils
- Poland (20):
  - NZOZ Specjalistyczny Osrodek Dermatologiczny DERMAL s.c., Bialystok
  - DERMAPOLIS Medical Dermatology Center, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - MCBK, Grodzisk Mazowiecki
  - Care Clinic Centrum Medyczne, Katowice
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Medyczne Promed, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej "DERMED" Centrum Medyczne, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Gabinety Lekarskie Rivermed, Poznan
  - Spolka Cywilna Andrzej Krolicki, Tomasz Kochanowski, ,,Laser Clinic", Szczecin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Medycyna Kliniczna, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej, Wroclaw
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Kliniczny Oddzial Chorob Wewnetrznych, Dermatologii i Alergologii, Zabrze
- Slovakia (6):
  - SUMMIT CLINICAL RESEARCH, s.r.o., Bratislava
  - SKINKLINIK s.r.o, Bratislava
  - BeneDerma s.r.o., Bratislava
  - Derma therapy spol. s.r.o., Bratislava
  - Dermatovenerologicka ambulancia, Nové Zámky
  - SANARE spol.s.r.o., Svidník
- South Korea (5):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Centro de Especialidades Mollabao (Area Sanitaria de Pontevedra e O Salnes), Pontevedra
  - Hospital de Montecelo, Pontevedra
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei, Taiwan (r.o.c)
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Simpson EL, Silverberg JI, Geng B, Carrascosa JM, Bieber T, Brunner PM, Staumont-Salle D, Ji C, Biswas P, Feeney C, Hernandez-Martin I, Rebollo Laserna FJ, Koppensteiner H. Do Allergic Comorbidities Alter the Efficacy and Safety of Abrocitinib or Dupilumab in Patients with Moderate-to-Severe Atopic Dermatitis? Dermatol Ther (Heidelb). 2025 Nov;15(11):3391-3407. doi: 10.1007/s13555-025-01516-w. Epub 2025 Sep 23. PMID 40987931
- [Derived] Silverberg JI, Simpson EL, Pink AE, Weidinger S, Chan G, Biswas P, Clibborn C, Guler E. Switching from Dupilumab to Abrocitinib in Patients With Moderate-to-Severe Atopic Dermatitis: A Post Hoc Analysis of Efficacy After Treatment With Dupilumab in JADE DARE. Dermatol Ther (Heidelb). 2025 Feb;15(2):367-380. doi: 10.1007/s13555-024-01320-y. Epub 2025 Feb 4. PMID 39903335
- [Derived] Reich K, Thyssen JP, Blauvelt A, Eyerich K, Soong W, Rice ZP, Hong HC, Katoh N, Valenzuela F, DiBonaventura M, Bratt TA, Zhang F, Clibborn C, Rojo R, Valdez H, Kerkmann U. Comparing how well abrocitinib and dupilumab treat atopic dermatitis signs and symptoms: a plain language summary. Immunotherapy. 2023 Sep;15(13):975-980. doi: 10.2217/imt-2022-0306. Epub 2023 May 31. PMID 37254941
- [Derived] Reich K, Thyssen JP, Blauvelt A, Eyerich K, Soong W, Rice ZP, Hong HC, Katoh N, Valenzuela F, DiBonaventura M, Bratt TA, Zhang F, Clibborn C, Rojo R, Valdez H, Kerkmann U. Efficacy and safety of abrocitinib versus dupilumab in adults with moderate-to-severe atopic dermatitis: a randomised, double-blind, multicentre phase 3 trial. Lancet. 2022 Jul 23;400(10348):273-282. doi: 10.1016/S0140-6736(22)01199-0. PMID 35871814
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, double-dummy, active-controlled study in adult participants with moderate to severe atopic dermatitis. The study was conducted across 143 sites in 15 countries.
Pre-assignment Details: A total of 940 participants were screened, of which 213 were screen failures and were not enrolled. 727 participants were enrolled in the study and assigned to a study intervention.
Groups:
- Abrocitinib 200 mg QD: Participants were administered abrocitinib 200 mg (2 x 100 mg) oral tablets once daily (QD) from Day 1 to Week 26 along with dupilumab-matching placebo administered as a subcutaneous injection once every 2 weeks (Q2W) until Week 24. Participants were followed for up to 4 weeks post last dose of study intervention.
- Dupilumab 300 mg Q2W: Participants were administered dupilumab 300 mg as a subcutaneous injection Q2W until Week 24 along with abrocitinib-matching placebo oral tablets administered once daily from Day 1 to Week 26. Participants were followed for up to 4 weeks post last dose of study intervention.
Period: Overall Study
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Started | 362 | 365
Completed | 327 | 334
Not Completed | 35 | 31
Not completed — Other | 3 | 4
Not completed — Medication Error Without Associated Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 2 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Death | 2 | 0
Not completed — Adverse Event | 10 | 9

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set comprised of all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W | Total
Number analyzed (Participants) | 362 | 365 | 727
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (14.6) | 35.5 (13.3) | 36.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 161 | 330
  Male | 193 | 204 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 27 | 57
  Not Hispanic or Latino | 331 | 337 | 668
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 62 | 83 | 145
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 26 | 51
  White | 269 | 248 | 517
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 4 Points Improvement in Peak Pruritus Numerical Rating Scale (PP-NRS4) From Baseline at Week 2
Description: The severity of itch (pruritus) due to atopic dermatitis (AD) was assessed using the PP-NRS, a validated horizontal NRS. Participants were asked to assess their worst itching due to AD over the past 24 hours on an NRS with scale ranging from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Week 2
Population: Full Analysis Set (FAS) comprised of all randomized participants who received at least one dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 357 | 364
Percentage of participants | 48.2 [43.0 to 53.4] | 25.5 [21.1 to 30.0]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) method adjusted by baseline disease severity; Estimate of difference = 22.6, 95% CI 2-sided [15.8 to 29.5] — The estimate and confidence interval (CI) for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions

2. Primary Outcome: Percentage of Participants Achieving >= 90% Improvement From Baseline in Eczema Area and Severity Index (EASI-90) Response at Week 4
Description: EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Time Frame: Week 4
Population: FAS comprised of all randomized participants who received at least one dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 354 | 364
Percentage of participants | 28.5 [23.8 to 33.2] | 14.6 [10.9 to 18.2]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — CMH method adjusted by baseline disease severity; Estimate of difference = 14.1, 95% CI 2-sided [8.2 to 20.0] — The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions

3. Secondary Outcome: Percentage of Participants Achieving EASI-90 Response at Week 16
Description: EASI quantifies severity of AD based on severity of lesion clinical signs and % of BSA affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 357 | 360
Percentage of participants | 54.3 [49.2 to 59.5] | 41.9 [36.8 to 47.0]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — CMH method adjusted by baseline disease severity; Estimate of difference = 12.5, 95% CI 2-sided [5.3 to 19.7] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving EASI-90 Response at Weeks 2, 8, 12, 20 and 26
Description: as for outcome 3
Time Frame: Week 2, 8, 12, 20 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention. Here, 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Week 2: number analyzed (Participants) | 361 | 362
  Week 2 | 11.6 [8.3 to 14.9] | 7.2 [4.5 to 9.8]
  Week 8: number analyzed (Participants) | 355 | 362
  Week 8 | 45.4 [40.2 to 50.5] | 25.4 [20.9 to 29.9]
  Week 12: number analyzed (Participants) | 359 | 363
  Week 12 | 47.6 [42.5 to 52.8] | 33.6 [28.7 to 38.5]
  Week 20: number analyzed (Participants) | 356 | 363
  Week 20 | 58.4 [53.3 to 63.5] | 45.7 [40.6 to 50.9]
  Week 26: number analyzed (Participants) | 348 | 361
  Week 26 | 54.6 [49.4 to 59.8] | 47.6 [42.5 to 52.8]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 4.5, 95% CI 2-sided [0.2 to 8.7] — Week 2. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 20.0, 95% CI 2-sided [13.2 to 26.9] — Week 8. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 14.0, 95% CI 2-sided [6.9 to 21.1] — Week 12. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 12.7, 95% CI 2-sided [5.5 to 20.0] — Week 20. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 6.9, 95% CI 2-sided [-0.4 to 14.3] — Week 26. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions

5. Secondary Outcome: Percentage of Participants Achieving >= 75% Improvement From Baseline in EASI (EASI-75) Response at Weeks 2, 4, 8, 12, 16, 20 and 26
Description: as for outcome 3
Time Frame: Week 2, 4, 8, 12, 16, 20 and 26
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Week 2: number analyzed (Participants) | 361 | 362
  Week 2 | 29.4 [24.7 to 34.1] | 21.3 [17.1 to 25.5]
  Week 4: number analyzed (Participants) | 354 | 364
  Week 4 | 57.6 [52.5 to 62.8] | 36.8 [31.9 to 41.8]
  Week 8: number analyzed (Participants) | 355 | 362
  Week 8 | 71.0 [66.3 to 75.7] | 52.8 [47.6 to 57.9]
  Week 12: number analyzed (Participants) | 359 | 363
  Week 12 | 76.3 [71.9 to 80.7] | 61.4 [56.4 to 66.4]
  Week 16: number analyzed (Participants) | 357 | 360
  Week 16 | 77.3 [73.0 to 81.7] | 67.8 [63.0 to 72.6]
  Week 20: number analyzed (Participants) | 356 | 363
  Week 20 | 76.1 [71.7 to 80.6] | 71.1 [66.4 to 75.7]
  Week 26: number analyzed (Participants) | 348 | 361
  Week 26 | 73.0 [68.3 to 77.7] | 72.3 [67.7 to 76.9]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 8.1, 95% CI 2-sided [1.8 to 14.4] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 20.9, 95% CI 2-sided [13.8 to 28.0] — Week 4. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 18.4, 95% CI 2-sided [11.4 to 25.3] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 14.9, 95% CI 2-sided [8.2 to 21.5] — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 9.5, 95% CI 2-sided [3.0 to 16.0] — Week 16. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 5.0, 95% CI 2-sided [-1.4 to 11.5] — [estimate comment as in outcome 4, analysis 4]
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 0.7, 95% CI 2-sided [-5.9 to 7.2] — [estimate comment as in outcome 4, analysis 5]

6. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' and >=2 Points Improvement From Baseline up to Week 26
Description: IGA assessed severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, except any residual discoloration (post-inflammatory hyperpigmentation and/or hypopigmentation); 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting.
Time Frame: Week 2, 4, 8, 12, 16, 20 and 26
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Week 2: number analyzed (Participants) | 361 | 362
  Week 2 | 14.4 [10.8 to 18.0] | 7.2 [4.5 to 9.8]
  Week 4: number analyzed (Participants) | 353 | 364
  Week 4 | 38.0 [32.9 to 43.0] | 17.6 [13.7 to 21.5]
  Week 8: number analyzed (Participants) | 355 | 362
  Week 8 | 50.1 [44.9 to 55.3] | 30.9 [26.2 to 35.7]
  Week 12: number analyzed (Participants) | 359 | 364
  Week 12 | 51.8 [46.6 to 57.0] | 36.0 [31.1 to 40.9]
  Week 16: number analyzed (Participants) | 358 | 360
  Week 16 | 55.3 [50.2 to 60.5] | 42.5 [37.4 to 47.6]
  Week 20: number analyzed (Participants) | 355 | 364
  Week 20 | 60.0 [54.9 to 65.1] | 50.8 [45.7 to 56.0]
  Week 26: number analyzed (Participants) | 347 | 362
  Week 26 | 55.6 [50.4 to 60.8] | 51.1 [46.0 to 56.3]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 7.3, 95% CI 2-sided [2.8 to 11.7] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 20.6, 95% CI 2-sided [14.3 to 26.9] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 19.5, 95% CI 2-sided [12.5 to 26.4] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 15.8, 95% CI 2-sided [8.7 to 23.0] — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 13.0, 95% CI 2-sided [5.9 to 20.2] — [estimate comment as in outcome 5, analysis 5]
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 9.2, 95% CI 2-sided [2.0 to 16.4] — [estimate comment as in outcome 4, analysis 4]
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 4.5, 95% CI 2-sided [-2.8 to 11.8] — [estimate comment as in outcome 4, analysis 5]

7. Secondary Outcome: Percentage of Participants Achieving PP-NRS4 From Baseline at Days 2 to 15
Description: The severity of itch (pruritus) due to AD was assessed using the PP-NRS, a validated horizontal NRS. Participants were asked to assess their worst itching due to AD over the past 24 hours on an NRS with scale ranging from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Day 2: number analyzed (Participants) | 319 | 317
  Day 2 | 11.0 [7.5 to 14.4] | 3.8 [1.7 to 5.9]
  Day 3: number analyzed (Participants) | 345 | 350
  Day 3 | 15.1 [11.3 to 18.8] | 8.6 [5.6 to 11.5]
  Day 4: number analyzed (Participants) | 349 | 356
  Day 4 | 22.1 [17.7 to 26.4] | 10.7 [7.5 to 13.9]
  Day 5: number analyzed (Participants) | 352 | 353
  Day 5 | 26.4 [21.8 to 31.0] | 11.9 [8.5 to 15.3]
  Day 6: number analyzed (Participants) | 348 | 348
  Day 6 | 28.4 [23.7 to 33.2] | 15.5 [11.7 to 19.3]
  Day 7: number analyzed (Participants) | 347 | 355
  Day 7 | 33.1 [28.2 to 38.1] | 13.2 [9.7 to 16.8]
  Day 8: number analyzed (Participants) | 353 | 347
  Day 8 | 36.3 [31.2 to 41.3] | 14.1 [10.5 to 17.8]
  Day 9: number analyzed (Participants) | 348 | 350
  Day 9 | 38.5 [33.4 to 43.6] | 16.9 [12.9 to 20.8]
  Day 10: number analyzed (Participants) | 345 | 353
  Day 10 | 40.0 [34.8 to 45.2] | 18.7 [14.6 to 22.8]
  Day 11: number analyzed (Participants) | 349 | 347
  Day 11 | 40.1 [35.0 to 45.3] | 20.2 [16.0 to 24.4]
  Day 12: number analyzed (Participants) | 347 | 351
  Day 12 | 41.5 [36.3 to 46.7] | 20.2 [16.0 to 24.4]
  Day 13: number analyzed (Participants) | 348 | 354
  Day 13 | 44.0 [38.8 to 49.2] | 21.5 [17.2 to 25.7]
  Day 14: number analyzed (Participants) | 347 | 354
  Day 14 | 45.5 [40.3 to 50.8] | 23.2 [18.8 to 27.6]
  Day 15: number analyzed (Participants) | 350 | 359
  Day 15 | 48.6 [43.3 to 53.8] | 25.6 [21.1 to 30.1]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 7.1, 95% CI 2-sided [3.1 to 11.1] — Day 2. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 6.5, 95% CI 2-sided [1.7 to 11.3] — Day 3. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 11.4, 95% CI 2-sided [6.0 to 16.8] — Day 4. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 14.5, 95% CI 2-sided [8.8 to 20.3] — Day 5. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 12.9, 95% CI 2-sided [6.9 to 19.0] — Day 6. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 19.9, 95% CI 2-sided [13.8 to 26.0] — Day 7. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 22.1, 95% CI 2-sided [15.9 to 28.3] — Day 8. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 8: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 21.7, 95% CI 2-sided [15.2 to 28.1] — Day 9. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 9: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of other = 21.3, 95% CI 2-sided [14.7 to 27.9] — Day 10. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 10: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 20.0, 95% CI 2-sided [13.3 to 26.6] — Day 11. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 11: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 21.3, 95% CI 2-sided [14.6 to 27.9] — Day 12. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 12: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 22.5, 95% CI 2-sided [15.8 to 29.2] — Day 13. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 13: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 22.4, 95% CI 2-sided [15.6 to 29.2] — Day 14. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions
Statistical Analysis 14: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 22.9, 95% CI 2-sided [16.0 to 29.9] — Day 15. The estimate and CI for difference were calculated based on the weighted average of difference by disease severity group using the normal approximation of binomial proportions

8. Secondary Outcome: Percentage of Participants Achieving PP-NRS4 From Baseline at Week 4, 8, 12, 16, 20 and 26
Description: as for outcome 7
Time Frame: Week 4, 8, 12, 16, 20 and 26
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Week 4: number analyzed (Participants) | 356 | 363
  Week 4 | 58.1 [53.0 to 63.3] | 40.8 [35.7 to 45.8]
  Week 8: number analyzed (Participants) | 357 | 364
  Week 8 | 65.8 [60.9 to 70.7] | 52.7 [47.6 to 57.9]
  Week 12: number analyzed (Participants) | 356 | 364
  Week 12 | 66.0 [61.1 to 70.9] | 61.5 [56.5 to 66.5]
  Week 16: number analyzed (Participants) | 357 | 363
  Week 16 | 67.2 [62.4 to 72.1] | 63.6 [58.7 to 68.6]
  Week 20: number analyzed (Participants) | 357 | 364
  Week 20 | 65.3 [60.3 to 70.2] | 63.2 [58.2 to 68.1]
  Week 26: number analyzed (Participants) | 354 | 363
  Week 26 | 68.1 [63.2 to 72.9] | 63.1 [58.1 to 68.0]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 17.3, 95% CI 2-sided [10.1 to 24.5] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 13.0, 95% CI 2-sided [6.0 to 20.1] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 4.4, 95% CI 2-sided [-2.5 to 11.4] — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 3.6, 95% CI 2-sided [-3.4 to 10.5] — [estimate comment as in outcome 5, analysis 5]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 2.0, 95% CI 2-sided [-4.9 to 9.0] — [estimate comment as in outcome 4, analysis 4]
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 5.0, 95% CI 2-sided [-1.9 to 11.9] — [estimate comment as in outcome 4, analysis 5]

9. Secondary Outcome: Time to Achieve >=4 Points Improvement in Peak Pruritus Numerical Rating Scale (PP-NRS4)
Description: as for outcome 7
Time Frame: Baseline (Day 1) up to Week 30
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 313 | 303
Days | 11.0 [9.0 to 14.0] | 25.0 [21.0 to 30.0]

10. Secondary Outcome: Percent Change From Baseline in the Percentage (%) Body Surface Area (BSA) Affected at Week 2, 4, 8, 12, 16, 20 and 26
Description: The extent (%) to which a body region was involved with AD was determined using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin/genitals) and lower limbs (including buttocks). Total number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual was derived as sum of % BSA across all 4 body regions and ranged from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline (Day 1), Week 2, 4, 8, 12, 16, 20 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percent change
  Week 2 | -42.7 [-46.0 to -39.4] | -33.4 [-36.7 to -30.0]
  Week 4 | -62.0 [-65.5 to -58.5] | -49.5 [-53.0 to -46.1]
  Week 8 | -74.0 [-77.2 to -70.7] | -62.8 [-66.0 to -59.7]
  Week 12 | -78.8 [-81.9 to -75.7] | -69.4 [-72.5 to -66.4]
  Week 16 | -80.6 [-83.5 to -77.8] | -73.7 [-76.5 to -70.9]
  Week 20 | -82.2 [-84.8 to -79.6] | -76.9 [-79.5 to -74.3]
  Week 26 | -82.3 [-85.0 to -79.6] | -79.0 [-81.6 to -76.3]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -9.3, 95% CI 2-sided [-14.0 to -4.6] — Week 2. Analysis was performed using Mixed Model Repeated Measure (MMRM) with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -12.5, 95% CI 2-sided [-17.4 to -7.6] — Week 4. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -11.1, 95% CI 2-sided [-15.6 to -6.6] — Week 8. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -9.4, 95% CI 2-sided [-13.7 to -5.1] — Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -6.9, 95% CI 2-sided [-10.9 to -2.9] — Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -5.3, 95% CI 2-sided [-9.0 to -1.7] — Week 20. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -3.4, 95% CI 2-sided [-7.1 to 0.4] — Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix

11. Secondary Outcome: Percent Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Total Score at Week 2, 4, 8, 12, 16, 20 and 26
Description: SCORAD is a scoring index for AD which combined extent (A), severity (B) and subjective symptoms (C). For A, a rule of 9 was used to calculate BSA affected by AD as % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; genitals 1%. Score of each body region was added to determine A (range: 0-100). B: severity of each sign (erythema; edema/papulation; oozing/crusting; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2), severe (3); severity scores were added to give B (range: 0-18). C: pruritus and sleep loss, each of these 2 were scored by participant/caregiver using visual analog scale (VAS) where, 0=no itch/no sleep loss and 10=worst imaginable itch/sleep loss, higher scores=worse symptoms. Scores for itch and sleep loss were added to give 'C' (range: 0-20). SCORAD total score was calculated as: A/5+7*B/2+C; range (0-103); higher values=worse outcome.
Time Frame: Baseline (Day 1), Week 2, 4, 8, 12, 16, 20 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percent change
  Week 2 | -44.5 [-47.0 to -42.1] | -33.5 [-35.9 to -31.0]
  Week 4 | -59.6 [-61.9 to -57.3] | -46.8 [-49.1 to -44.5]
  Week 8 | -65.8 [-68.2 to -63.4] | -55.6 [-58.0 to -53.3]
  Week 12 | -67.9 [-70.2 to -65.6] | -60.6 [-62.9 to -58.3]
  Week 16 | -70.6 [-72.8 to -68.3] | -64.4 [-66.7 to -62.2]
  Week 20 | -71.8 [-74.1 to -69.4] | -66.8 [-69.1 to -64.5]
  Week 26 | -71.5 [-73.9 to -69.1] | -68.2 [-70.6 to -65.9]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -11.0, 95% CI 2-sided [-14.5 to -7.6] — Week 2. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -12.8, 95% CI 2-sided [-16.0 to -9.5] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -10.2, 95% CI 2-sided [-13.6 to -6.8] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -7.3, 95% CI 2-sided [-10.5 to -4.1] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -6.1, 95% CI 2-sided [-9.3 to -3.0] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -4.9, 95% CI 2-sided [-8.2 to -1.7] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -3.3, 95% CI 2-sided [-6.6 to 0.1] — [estimate comment as in outcome 10, analysis 7]

12. Secondary Outcome: Change From Baseline in Total Anxiety Score Measured Using the Hospital Anxiety and Depression Scale (HADS) at Week 12,16 and 26
Description: HADS was a validated 14-item questionnaire to assess states of anxiety and depression over the past week. HADS consisted of 2 subscales: HADS-Anxiety (HADS-A) scale and HADS-Depression (HADS-D) scale, each of which comprised of 7 items. Each item was rated on a 4-point scale, with scores ranging from 0 to 3, where higher scores indicated more anxiety/depression symptoms. HADS-A assessed state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-A total score was calculated as the sum of all 7 items with score ranging from 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicated greater severity of anxiety.
Time Frame: Baseline (Day 1), Week 12, 16 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Units on a scale
  Week 12 | -0.8 [-1.1 to -0.5] | -0.8 [-1.1 to -0.6]
  Week 16 | -1.1 [-1.3 to -0.8] | -1.2 [-1.4 to -0.9]
  Week 26 | -1.1 [-1.4 to -0.7] | -1.2 [-1.5 to -0.9]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.4] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.3 to 0.5] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.3 to 0.6] — [estimate comment as in outcome 10, analysis 7]

13. Secondary Outcome: Change From Baseline in Total Depression Score Measured Using the HADS at Week 12,16 and 26
Description: HADS was a validated 14-item questionnaire to assess states of anxiety and depression over the past week. HADS consisted of 2 subscales: HADS-A scale and HADS-D scale, each of which comprised of 7 items. Each item was rated on a 4-point scale, with scores ranging from 0 to 3, where higher scores indicated more anxiety/depression symptoms. HADS-D assessed the state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-D: total score was calculated as the sum of all 7 items with score ranging from 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicated greater severity of depression symptoms.
Time Frame: Baseline (Day 1), Week 12, 16 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Units on a scale
  Week 12 | -0.7 [-1.0 to -0.5] | -0.7 [-1.0 to -0.5]
  Week 16 | -0.8 [-1.0 to -0.5] | -0.9 [-1.1 to -0.7]
  Week 26 | -0.8 [-1.0 to -0.5] | -1.0 [-1.3 to -0.8]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.0, 95% CI 2-sided [-0.3 to 0.3] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.5] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.2, 95% CI 2-sided [-0.1 to 0.6] — [estimate comment as in outcome 10, analysis 7]

14. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 2, 12, 16, 20 and 26
Description: DLQI is a 10-item questionnaire that measured the impact of skin disease. Each question was evaluated on a 4-point scale (range 0 to 3) where, 0 = not at all, 1= a little, 2= a lot, 3= very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score, ranging from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline (Day 1), Week 2, 12, 16, 20 and 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 361 | 363
Units on a scale
  Week 2 | -8.6 [-9.1 to -8.2] | -6.7 [-7.1 to -6.2]
  Week 12 | -10.7 [-11.1 to -10.2] | -9.7 [-10.1 to -9.3]
  Week 16 | -10.8 [-11.2 to -10.4] | -10.0 [-10.5 to -9.6]
  Week 20 | -10.8 [-11.2 to -10.3] | -10.1 [-10.6 to -9.7]
  Week 26 | -10.3 [-10.8 to -9.9] | -10.0 [-10.5 to -9.6]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.0, 95% CI 2-sided [-2.6 to -1.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.0, 95% CI 2-sided [-1.6 to -0.4] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.8, 95% CI 2-sided [-1.4 to -0.2] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.6, 95% CI 2-sided [-1.2 to 0.0] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.3, 95% CI 2-sided [-1.0 to 0.4] — [estimate comment as in outcome 10, analysis 7]

15. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension 5-Level (EQ-5D-5L) Visual Analog Scale (VAS) Score at Week 12, 16 and 26
Description: The EQ-5D-5L is a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score. There were two components to the EQ-5D-5L: a five-item health state profile that assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a VAS that measured health state. EQ-5D VAS was used to record participant's rating for his/her current health-related quality of life state on a vertical VAS with scores ranging from 0 to 100, where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline (Day 1), Week 12, 16 and 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 364
Units on a scale
  Week 12 | 12.370 [10.917 to 13.822] | 11.552 [10.123 to 12.981]
  Week 16 | 12.567 [11.015 to 14.118] | 10.474 [8.951 to 11.997]
  Week 26 | 13.484 [11.982 to 14.985] | 14.300 [12.836 to 15.764]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.818, 95% CI 2-sided [-1.220 to 2.856] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 2.093, 95% CI 2-sided [-0.081 to 4.267] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.816, 95% CI 2-sided [-2.914 to 1.281] — [estimate comment as in outcome 10, analysis 7]

16. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Total Score at Week 12, 16 and 26
Description: POEM was a 7-item participant reported outcome measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item was scored as: no days=0, 1-2 days=1, 3-4 days=2, 5-6 days=3 and every day=4. The item scores were added to provide a total score ranging from 0 to 28, where higher score indicated greater severity.
Time Frame: Baseline (Day 1), Week 12, 16 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Units on a scale
  Week 12 | -14.2 [-14.9 to -13.6] | -12.6 [-13.3 to -12.0]
  Week 16 | -14.2 [-14.8 to -13.6] | -12.8 [-13.4 to -12.2]
  Week 26 | -13.8 [-14.5 to -13.1] | -13.4 [-14.0 to -12.7]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.6, 95% CI 2-sided [-2.5 to -0.7] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.4, 95% CI 2-sided [-2.2 to -0.5] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.4, 95% CI 2-sided [-1.3 to 0.5] — [estimate comment as in outcome 10, analysis 7]

17. Secondary Outcome: Change From Baseline in Medical Outcomes Study - Sleep Scale (MOS-Sleep Scale) at Week 12, 16 and 26
Description: The MOS Sleep Scale is a 12-item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, short of breath or headache, adequacy of sleep, somnolence, sleep problems index I and sleep problems index II). An additional single item assessed quantity of sleep. Each of the sleep domains were scored on a range of 0 to 100, and higher scores indicated worse outcomes. The quantity of sleep scores ranged from 0 to 24 (number of hours slept). Change from baseline scores for each individual sleep domain and quantity of sleep are reported in this outcome measure.
Time Frame: Baseline (Day 1), Week 12, 16 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Units on a scale
  Quantity Hours Slept Score: Week 12 | 0.7 [0.5 to 0.9] | 0.5 [0.2 to 0.7]
  Quantity Hours Slept Score: Week 16 | 0.6 [0.3 to 0.8] | 0.5 [0.3 to 0.7]
  Quantity Hours Slept Score: Week 26 | 0.5 [0.3 to 0.7] | 0.4 [0.2 to 0.6]
  Short of Breath or Headache score: Week 12 | -0.7 [-2.2 to 0.9] | -1.9 [-3.4 to -0.4]
  Short of Breath or Headache score: Week 16 | -1.2 [-2.7 to 0.3] | -1.3 [-2.8 to 0.2]
  Short of Breath or Headache score: Week 26 | -2.0 [-3.5 to -0.6] | -2.6 [-4.0 to -1.2]
  Snoring Score: Week 12 | -5.3 [-7.0 to -3.6] | -3.5 [-5.2 to -1.8]
  Snoring Score: Week 16 | -4.9 [-6.6 to -3.1] | -4.0 [-5.7 to -2.3]
  Snoring Score: Week 26 | -3.9 [-5.7 to -2.0] | -4.7 [-6.5 to -2.9]
  Sleep Disturbance Score: Week 12 | -20.5 [-22.3 to -18.8] | -16.4 [-18.1 to -14.7]
  Sleep Disturbance Score: Week 16 | -21.5 [-23.2 to -19.7] | -17.7 [-19.4 to -16.0]
  Sleep Disturbance Score: Week 26 | -21.2 [-23.0 to -19.5] | -19.5 [-21.2 to -17.8]
  Sleep Adequacy Score: Week 12 | 13.9 [12.1 to 15.8] | 12.9 [11.1 to 14.7]
  Sleep Adequacy Score: Week 16 | 15.7 [13.9 to 17.4] | 12.7 [11.0 to 14.5]
  Sleep Adequacy Score: Week 26 | 14.0 [12.1 to 15.8] | 13.2 [11.4 to 15.1]
  Sleep Somnolence Score: Week 12 | -7.7 [-9.1 to -6.2] | -6.9 [-8.3 to -5.5]
  Sleep Somnolence Score: Week 16 | -9.8 [-11.3 to -8.4] | -7.4 [-8.8 to -6.0]
  Sleep Somnolence Score: Week 26 | -9.9 [-11.3 to -8.5] | -7.6 [-9.0 to -6.2]
  Sleep Problems Index I Score: Week 12 | -12.1 [-13.4 to -10.8] | -10.9 [-12.2 to -9.6]
  Sleep Problems Index I Score: Week 16 | -13.3 [-14.5 to -12.0] | -11.0 [-12.2 to -9.8]
  Sleep Problems Index I Score: Week 26 | -12.9 [-14.2 to -11.7] | -12.1 [-13.3 to -10.9]
  Sleep Problems Index II Score: Week 12 | -14.4 [-15.7 to -13.1] | -12.2 [-13.5 to -10.9]
  Sleep Problems Index II Score: Week 16 | -15.7 [-17.0 to -14.4] | -12.8 [-14.0 to -11.5]
  Sleep Problems Index II Score: Week 26 | -15.4 [-16.7 to -14.1] | -14.0 [-15.2 to -12.7]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.2, 95% CI 2-sided [-0.1 to 0.6] — Quantity of hours slept: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.4] — Quantity of hours slept: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.4] — Quantity of hours slept: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 1.2, 95% CI 2-sided [-0.9 to 3.4] — Short of Breath or Headache score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-2.0 to 2.2] — Short of Breath or Headache score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 6: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.6, 95% CI 2-sided [-1.5 to 2.6] — Short of Breath or Headache score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 7: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.8, 95% CI 2-sided [-4.2 to 0.5] — Snoring score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 8: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.9, 95% CI 2-sided [-3.3 to 1.5] — Snoring score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 9: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.8, 95% CI 2-sided [-1.7 to 3.4] — Snoring score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 10: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -4.1, 95% CI 2-sided [-6.6 to -1.6] — Sleep disturbance score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 11: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -3.8, 95% CI 2-sided [-6.2 to -1.4] — Sleep disturbance score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 12: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.7, 95% CI 2-sided [-4.1 to 0.7] — Sleep disturbance score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 13: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 1.0, 95% CI 2-sided [-1.6 to 3.6] — Sleep adequacy score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 14: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 2.9, 95% CI 2-sided [0.4 to 5.4] — Sleep adequacy score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 15: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = 0.7, 95% CI 2-sided [-1.9 to 3.4] — Sleep adequacy score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 16: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.8, 95% CI 2-sided [-2.8 to 1.3] — Sleep somnolence score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 17: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.4, 95% CI 2-sided [-4.4 to -0.4] — Sleep somnolence score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 18: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.3, 95% CI 2-sided [-4.3 to -0.3] — Sleep somnolence score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 19: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.2, 95% CI 2-sided [-3.0 to 0.7] — Sleep Problems Index I score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 20: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.3, 95% CI 2-sided [-4.0 to -0.5] — Sleep Problems Index I score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 21: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.8, 95% CI 2-sided [-2.5 to 0.9] — Sleep Problems Index I score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 22: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.2, 95% CI 2-sided [-4.0 to -0.3] — Sleep Problems Index II score: Week 12. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 23: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -2.9, 95% CI 2-sided [-4.8 to -1.1] — Sleep Problems Index II score: Week 16. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix
Statistical Analysis 24: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.4, 95% CI 2-sided [-3.2 to 0.4] — Sleep Problems Index II score: Week 26. Analysis was performed using MMRM with fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, baseline value and an unstructured covariance matrix

18. Secondary Outcome: Change From Baseline in Skin Pain NRS at Week 2, 12, 16, 20 and 26
Description: The skin pain NRS was a participant reported outcome where participants were asked to rate the "worst skin pain" in the past 24 hours on a 11-point scale from 0=no skin pain to 10=worst skin pain imaginable. Higher scores indicated worse pain.
Time Frame: Baseline (Day 1), Week 2, 12, 16, 20 and 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Units on a scale
  Week 2 | -3.7 [-3.9 to -3.4] | -2.6 [-2.8 to -2.3]
  Week 12 | -4.5 [-4.7 to -4.2] | -4.0 [-4.3 to -3.8]
  Week 16 | -4.4 [-4.7 to -4.2] | -4.2 [-4.4 to -4.0]
  Week 20 | -4.8 [-5.0 to -4.5] | -4.5 [-4.7 to -4.2]
  Week 26 | -4.5 [-4.8 to -4.3] | -4.3 [-4.6 to -4.1]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -1.1, 95% CI 2-sided [-1.5 to -0.8] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.4, 95% CI 2-sided [-0.8 to -0.1] — [estimate comment as in outcome 10, analysis 4]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.1] — [estimate comment as in outcome 10, analysis 5]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.3, 95% CI 2-sided [-0.6 to 0.0] — [estimate comment as in outcome 10, analysis 6]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Least square mean difference = -0.2, 95% CI 2-sided [-0.5 to 0.1] — [estimate comment as in outcome 10, analysis 7]

19. Secondary Outcome: Medicated Topical Background Therapy-free Days
Description: Medicated topical background therapy-free days was defined as number of days where a participant maintained a response of EASI-90 or greater without the use of medicated topical background therapy.
Time Frame: Day 1 up to Week 26
Population: FAS comprised of all randomized participants who received at least one dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Days | 51.4 [46.0 to 56.8] | 33.3 [27.9 to 38.7]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Analysis was performed using analysis of covariance (ANCOVA) model including treatment as a main effect and baseline disease severity as covariates; Test type: Other; Least square mean difference = 18.1, 95% CI 2-sided [10.5 to 25.7]

20. Secondary Outcome: Percentage of Participants Achieving >=4 Points Improvement From Baseline in DLQI at Week 2, 12, 16, 20 and 26
Description: DLQI was a 10-item questionnaire that measured the impact of skin disease. Each question was evaluated on a 4-point scale (range 0 to 3) where, 0 = not at all, 1= a little, 2= a lot, 3= very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Week 2, 12, 16, 20 and 26
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Percentage of participants
  Week 2: number analyzed (Participants) | 342 | 351
  Week 2 | 81.3 [77.2 to 85.4] | 67.5 [62.6 to 72.4]
  Week 12: number analyzed (Participants) | 343 | 350
  Week 12 | 85.4 [81.7 to 89.2] | 81.4 [77.4 to 85.5]
  Week 16: number analyzed (Participants) | 342 | 349
  Week 16 | 82.7 [78.7 to 86.8] | 84.2 [80.4 to 88.1]
  Week 20: number analyzed (Participants) | 341 | 350
  Week 20 | 81.8 [77.7 to 85.9] | 83.7 [79.8 to 87.6]
  Week 26: number analyzed (Participants) | 334 | 349
  Week 26 | 76.6 [72.1 to 81.2] | 80.8 [76.7 to 84.9]
Statistical Analysis 1: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 13.7, 95% CI 2-sided [7.3 to 20.1] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = 3.9, 95% CI 2-sided [-1.6 to 9.4] — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 3: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = -1.6, 95% CI 2-sided [-7.1 to 4.0] — [estimate comment as in outcome 5, analysis 5]
Statistical Analysis 4: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = -2.0, 95% CI 2-sided [-7.6 to 3.6] — [estimate comment as in outcome 4, analysis 4]
Statistical Analysis 5: Comparison: Abrocitinib 200 mg QD vs Dupilumab 300 mg Q2W; Test type: Other; Estimate of difference = -4.2, 95% CI 2-sided [-10.3 to 1.9] — [estimate comment as in outcome 4, analysis 5]

21. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a treatment-emergent adverse event (TEAE) if the event started on or after the first dosing day until 28 days post last dose of study drug. AEs included both serious and non-serious AEs.
Time Frame: From start of study intervention to 28 days post last dose of study intervention (Up to Week 30)
Population: Safety population comprised of all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Participants | 268 | 239

22. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs) and AEs Leading to Study Discontinuation
Description: An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; a congenital anomaly/birth defect and other important medical events.
Time Frame: From start of study intervention to 28 days post last dose of study intervention (Up to Week 30)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Participants
  SAEs | 6 | 6
  AEs Leading to Study Discontinuation | 12 | 9

23. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Meeting Pre-Defined Criteria
Description: The pre-defined criteria for laboratory parameters included: hemoglobin (<9 grams per deciliter or decreases to >=2 below baseline); platelets (<75*10^3 cells per millimeter cube [mm^3]); lymphocytes (<0.5*10^3 cells per mm^3); neutrophils (<1*10^3 cells per mm^3); aspartate aminotransferase and alanine aminotransferase (>3* upper limit of normal).
Time Frame: From start of study intervention to 28 days post last dose of study intervention (Up to Week 30)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Participants | 38 | 10

24. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs including temperature, systolic and diastolic blood pressure, and pulse rate were measured in a seated position after 5 minutes rest. Clinically significant change from baseline in vital signs were determined by the investigator.
Time Frame: From start of study intervention to 28 days post last dose of study intervention (Up to Week 30)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Participants | 0 | 0

25. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Data
Description: A single 12-lead ECG was performed after the participant has rested for at least 10 minutes quietly in the supine position. Clinically significant change from baseline in ECG data was determined by the investigator.
Time Frame: From start of study intervention to 28 days post last dose of study intervention (Up to Week 30)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 362 | 365
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study intervention up to 28 days after last dose of study intervention (Up to Week 30)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Abrocitinib 200 mg QD | Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 2/362 | 0/365
Serious Adverse Events (participants affected / at risk) | 6/362 | 6/365
Other Adverse Events (participants affected / at risk) | 203/362 | 144/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib 200 mg QD (N=362) | Dupilumab 300 mg Q2W (N=365)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib 200 mg QD (N=362) | Dupilumab 300 mg Q2W (N=365)
Diarrhoea (Gastrointestinal disorders) | 8 | 8
Nausea (Gastrointestinal disorders) | 70 | 8
Vomiting (Gastrointestinal disorders) | 11 | 6
Fatigue (General disorders) | 10 | 5
COVID-19 (Infections and infestations) | 14 | 12
Conjunctivitis (Infections and infestations) | 8 | 35
Folliculitis (Infections and infestations) | 12 | 3
Herpes simplex (Infections and infestations) | 12 | 5
Herpes zoster (Infections and infestations) | 9 | 2
Nasopharyngitis (Infections and infestations) | 14 | 12
Oral herpes (Infections and infestations) | 9 | 15
Upper respiratory tract infection (Infections and infestations) | 10 | 9
Urinary tract infection (Infections and infestations) | 8 | 7
Blood creatine phosphokinase increased (Investigations) | 14 | 13
Natural killer cell count decreased (Investigations) | 10 | 0
SARS-CoV-2 test positive (Investigations) | 15 | 13
Weight increased (Investigations) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Dizziness (Nervous system disorders) | 10 | 4
Headache (Nervous system disorders) | 47 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Acne (Skin and subcutaneous tissue disorders) | 46 | 10
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 17 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT04345367/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT04345367/SAP_001.pdf